CLINICAL TRIAL: NCT02079766
Title: 18F-AV-1451 and Florbetapir F 18 PET Imaging in Subjects With Repetitive Brain Trauma at High Risk for Chronic Traumatic Encephalopathy
Brief Title: 18F-AV-1451 and Florbetapir F 18 PET (Positron Emission Tomography) Imaging in Subjects at Risk for Chronic Traumatic Encephalopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 18F-AV-1451-A07
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Results first posted 2020-09-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Chronic Traumatic Encephalopathy
MeSH Terms: conditions — Chronic Traumatic Encephalopathy | interventions — florbetapir; 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Risk of CTE (Experimental): Flortaucipir PET scans in subjects at high risk of developing CTE (former National Football League players)
  Interventions: Drug: florbetapir F 18; Drug: Flortaucipir F18
- Control (Experimental): Flortaucipir PET scans in former non-contact athletes
  Interventions: Drug: florbetapir F 18; Drug: Flortaucipir F18

INTERVENTIONS:
Drug: florbetapir F 18 — 370 megabecquerel (MBq) IV single-dose
  Other Names: Amyvid; 18F-AV-45
Drug: Flortaucipir F18 — 370 megabecquerel (MBq) IV single-dose
  Other Names: T807; 18F-AV-1451; LY3191748

SUMMARY:
This study will explore the use of flortaucipir as a biomarker for chronic traumatic encephalopathy (CTE) and examine the relationship between clinical presentation and tau deposition.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects consented and currently enrolled in the Diagnosing and Evaluating Traumatic Encephalopathy Using Clinical Tests (DETECT) or the Long-Term Consequences of Repetitive Brain Injury in Athletes study protocols
* Can tolerate up to two PET imaging sessions
* Have the ability to provide informed consent for study procedures

Exclusion Criteria:

* Claustrophobia
* Current clinically significant cardiovascular disease or clinically significant abnormalities on screening ECG
* History of risk factors for Torsades de Pointes or are taking drugs known to cause QT-prolongation
* Current clinically significant infectious disease, endocrine or metabolic disease, pulmonary, renal or hepatic impairment, or cancer that the investigator believes would affect study participation or scan results
* Have had a non-study related radiopharmaceutical imaging or treatment within 7 days prior to study PET imaging sessions

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Chair — Avid Radiopharmaceuticals, Inc.
Locations (2):
- United States (2):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Boston University, Boston, Massachusetts

REFERENCES:
- [Result] Stern RA, Adler CH, Chen K, Navitsky M, Luo J, Dodick DW, Alosco ML, Tripodis Y, Goradia DD, Martin B, Mastroeni D, Fritts NG, Jarnagin J, Devous MD Sr, Mintun MA, Pontecorvo MJ, Shenton ME, Reiman EM. Tau Positron-Emission Tomography in Former National Football League Players. N Engl J Med. 2019 May 2;380(18):1716-1725. doi: 10.1056/NEJMoa1900757. Epub 2019 Apr 10. PMID 30969506

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited between June 2014 and October 2015 from the DETECT study (National Institutes of Health grant R01NS078337) and the Arizona Alzheimer's Consortium ("Long-Term Consequences of Repetitive Brain Injury in Athletes: A Longitudinal Study with Eventual Brain Donation")
Groups:
- High Risk of CTE: Subjects at high risk of developing CTE (chronic traumatic encephalopathy) - former National Football League players
- Controls: Former non-contact athletes
Period: Overall Study
Arm/Group | High Risk of CTE | Controls
Started | 30 | 11
Completed | 28 | 11
Not Completed | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Includes all subjects who received at least one dose of florbetapir or flortaucipir
Groups:
- High Risk of CTE: Subjects at high risk of developing CTE (former National Football League players)
- Total: Total of all reporting groups
Arm/Group | High Risk of CTE | Controls | Total
Number analyzed (Participants) | 29 | 11 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (8.27) | 57.4 (6.25) | 58.2 (7.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 29 | 11 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 29 | 11 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 14 | 1 | 15
  White | 14 | 10 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 11 | 40
MMSE [Mean (Standard Deviation); unit: units on a scale] — Mini-mental status exam is a 30-point questionnaire that is used to measure cognitive impairment. Scores range from 0 to 30 with lower scores representing greater levels of cognitive impairment.
  units on a scale | 27.2 (1.64) | 28.6 (0.92) | 27.6 (1.60)
Amyloid status [Count of Participants; unit: Participants] — Measured by flortaucipir PET scan visual read augmented with quantitative information Population: Only included subjects for which a florbetapir PET scan was available
  Participants
    number analyzed (Participants) | 28 | 11 | 39
    Amyloid positive | 3 | 0 | 3
    Amyloid Negative | 25 | 11 | 36

OUTCOME MEASURES:

1. Primary Outcome: Flortaucipir Visual Read as CTE Biomarker
Description: Flortaucipir uptake was rated visually by sponsor expert reader as 'No Uptake', 'Mild Uptake', 'Moderate Uptake', or 'Intense Uptake'.
Time Frame: Baseline scan
Population: All subjects who received a flortaucipir scan
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk of CTE | Controls
Number analyzed (Participants) | 28 | 11
Participants
  No Uptake | 23 | 11
  Mild Uptake | 5 | 0
  Moderate Uptake | 0 | 0
  Intense Uptake | 0 | 0
Statistical Analysis 1: Comparison: High Risk of CTE vs Controls; Evaluated the association between the overall brain uptake and the study group; Test type: Other; p = 0.2959, Fisher Exact — No adjustments for multiple comparisons or multiplicity were made for this study. No a priori threshold for significance was chosen

2. Primary Outcome: Relationship Between Clinical Presentation and Tau Deposition (Subjects at High Risk of CTE Only)
Description: The relationship between flortaucipir uptake and clinical presentation, as measured by the Mini-Mental State Examination (MMSE). Mini-mental status exam is a 30-point questionnaire that is used to measure cognitive impairment. Scores range from 0 to 30 with lower scores representing greater levels of cognitive impairment. Specified in statistical analysis plan to only be conducted in High Risk of CTE group.
Time Frame: baseline scan
Population: Only subjects at high risk for CTE were included in this analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | High Risk of CTE
Number analyzed (Participants) | 28
score on a scale
  No Uptake: number analyzed (Participants) | 23
  No Uptake | 27.348 [26.625 to 28.071]
  Mild Uptake: number analyzed (Participants) | 5
  Mild Uptake | 26.800 [25.249 to 28.351]
  Moderate Uptake: number analyzed (Participants) | 0
  Intense Uptake: number analyzed (Participants) | 0
Statistical Analysis 1: Comparison: High Risk of CTE; Measured differences in clinical presentation using MMSE between subjects with no visual flortaucipir uptake, and those with mild uptake; Test type: Other; p = 0.5163, ANOVA — [p-value comment as in outcome 1, analysis 1]; MMSE score as the response variable and flortaucipir uptake score (4 levels) as the fixed effect

ADVERSE EVENTS:
Time Frame: End of study for AE reporting was 48 hours after the last study drug administration.
Description: Adverse events (AEs) were collected at scan visits, regardless of attribution to study drug. AEs occurring after study drug administration, but outside that window were not recorded, unless considered attributable to either drug. Includes all subjects who received at least one dose of florbetapir or flortaucipir
Arm/Group | High Risk of CTE | Controls
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/11
Other Adverse Events (participants affected / at risk) | 11/29 | 5/11
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Risk of CTE (N=29) | Controls (N=11)
headache (Nervous system disorders) | 4 (4) | 2 (2)
nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
oral pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
dizziness (Nervous system disorders) | 0 (0) | 1 (1)
diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
fatigue (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less